CLINICAL TRIAL: NCT06319703
Title: IDEAL: Implementing an Effective Diabetes intervEntion Among Low-income Immigrants
Brief Title: Implementing an Effective Diabetes Intervention Among Low-Income Immigrants
Acronym: IDEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-00634
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: Mobile Health; mHealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSMES+CHW (IDEAL) (Experimental): Participants in this group will receive brief pre-recorded DSMES videos, which include both educational and Social Cognitive Theory-based behavioral content. Participants will receive 1 DSMES video via text message each week for a total of 24 weeks with each video lasting about 5 minutes in duration. In addition, they will also receive brief phone calls from CHWs every 2 weeks during the 24 weeks video program. During these calls, CHWs will assess whether participants need assistance on social determinants of health (SDOH) barriers. If needed, CHWs will link participants to available services within the community. CHWs will also provide assistance on navigating the complex health care systems and serve as an advocate for patients during doctor visits if needed.
  Interventions: Behavioral: Diabetes Self-Management Education and Support (DSMES) Videos; Behavioral: Community Health Worker Support (CHW)
- Wait-list control group (CONTROL) (No Intervention): Participants in this group will continue to receive the standard of usual care for their T2D at their doctor's office during the course of our study.

INTERVENTIONS:
Behavioral: Diabetes Self-Management Education and Support (DSMES) Videos — Text message-delivered video-based DSMES intervention.
  Arms: DSMES+CHW (IDEAL)
Behavioral: Community Health Worker Support (CHW) — Assess participants' SDOH barriers to Type 2 diabetes care and link them to available resources in the community.
  Arms: DSMES+CHW (IDEAL)

SUMMARY:
The goal of this IDEAL project is to examine the effectiveness and implementation process of the video-based Diabetes Self-Management Education and Support (DSMES) + community health worker (CHW) (hereafter: "IDEAL") intervention compared with a wait-list control group (hereafter: "CONTROL") to improve glycemic control among Chinese immigrants with Type 2 diabetes (T2D) in New York City (NYC). Participants will be randomized with equal allocation to one of the 2 groups. The IDEAL group will receive 1 DSMES brief video/week for 24 weeks delivered via text message. The CHW will assess participants' SDOH barriers to T2D care and link them to available resources in the community. The CONTROL group will continue to receive their usual care and at the end of the study, they will receive DSMES videos.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. self-identify as a Chinese immigrant;
2. be between 18-70 years old,
3. have a diagnosis of T2D in the medical record;
4. have had an appointment with a physician for routine T2D care within the past 12 months;
5. have a most recent HbA1c > or = 8%;
6. be willing to receive brief videos regarding T2D management, and
7. possess a smartphone or, if they do not have one, be willing and able to use a study smartphone.

Exclusion Criteria:

1. unable or unwilling to provide informed consent;
2. unable to participate meaningfully in the intervention (e.g., uncorrected sight and hearing impairment);
3. unwilling to accept randomization assignment;
4. is pregnant, plans to become pregnant in the next 6 months, or becomes pregnant during the study, or
5. is breastfeeding (e.g., they may have potential dietary restrictions).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-12-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C (HbA1c) Test Scores | Baseline, Month 6
  Scores expressed as a percentage of red blood cells that have sugar-coated hemoglobin.
  Patients with Type 2 Diabetes receive a HbA1c blood test at their doctors' office every 3-6 months as part of usual care; testing results will be abstracted from the medical record at the participant's health care facility to minimize participant burden.
Change in Hemoglobin A1C (HbA1c) Test Scores | Baseline, Month 12
  Scores expressed as a percentage of red blood cells that have sugar-coated hemoglobin.
  Patients with Type 2 Diabetes receive a HbA1c blood test at their doctors' office every 3-6 months as part of usual care; testing results will be abstracted from the medical record at the participant's health care facility to minimize participant burden.

SECONDARY OUTCOMES:
Stanford Self-Efficacy for Diabetes Scale Score | Baseline
  8-item self-assessment of participants' confidence level in performing specific self-management behaviors. Items are ranked on a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident).
  The score is the mean of the 8 items (Range: 1-10); higher scores indicate greater self-efficacy.
Stanford Self-Efficacy for Diabetes Scale Score | Month 6
  8-item self-assessment of participants' confidence level in performing specific self-management behaviors. Items are ranked on a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident).
  The score is the mean of the 8 items (Range: 1-10); higher scores indicate greater self-efficacy.
Stanford Self-Efficacy for Diabetes Scale Score | Month 12
  8-item self-assessment of participants' confidence level in performing specific self-management behaviors. Items are ranked on a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident).
  The score is the mean of the 8 items (Range: 1-10); higher scores indicate greater self-efficacy.
Summary of Diabetes Self-Care Activities (SDSCA) Score | Baseline
  11-item self-report questionnaire assessing participants' adherence to diabetes self-management behaviors. Participants select the number of days (0 to 7) in the past week they have performed the behavior.
  The result is an average score between 0 and 7; higher scores indicate better diabetes self-management behavior.
Summary of Diabetes Self-Care Activities (SDSCA) Score | Month 6
  11-item self-report questionnaire assessing participants' adherence to diabetes self-management behaviors. Participants select the number of days (0 to 7) in the past week they have performed the behavior.
  The result is an average score between 0 and 7; higher scores indicate better diabetes self-management behavior.
Summary of Diabetes Self-Care Activities (SDSCA) Score | Month 12
  11-item self-report questionnaire assessing participants' adherence to diabetes self-management behaviors. Participants select the number of days (0 to 7) in the past week they have performed the behavior.
  The result is an average score between 0 and 7; higher scores indicate better diabetes self-management behavior.
Starting the Conversation (STC) Diet Scale Score | Baseline
  8-item self-report questionnaire measuring dietary behaviors. Scores range from 0 to 16; higher scores indicate more dietary behaviors that are not consistent with health.
Starting the Conversation (STC) Diet Scale Score | Month 6
  8-item self-report questionnaire measuring dietary behaviors. Scores range from 0 to 16; higher scores indicate more dietary behaviors that are not consistent with health.
Starting the Conversation (STC) Diet Scale Score | Month 12
  8-item self-report questionnaire measuring dietary behaviors. Scores range from 0 to 16; higher scores indicate more dietary behaviors that are not consistent with health.
National Cancer Institute Dietary Screener Questionnaire Score | Baseline
  27-item self-assessment of frequency of consumption of selected foods and drinks over the past month.
  The scoring procedure converts responses to estimates of individual dietary intake for: Fruits and Vegetables (cup equivalents); Dairy (cup equivalents); Added Sugars (teaspoon equivalents); Whole Grains (ounce equivalents); Fiber (grams); and Calcium (milligrams). Higher scores indicate higher consumption of the food item.
National Cancer Institute Dietary Screener Questionnaire Score | Month 6
  27-item self-assessment of frequency of consumption of selected foods and drinks over the past month.
  The scoring procedure converts responses to estimates of individual dietary intake for: Fruits and Vegetables (cup equivalents); Dairy (cup equivalents); Added Sugars (teaspoon equivalents); Whole Grains (ounce equivalents); Fiber (grams); and Calcium (milligrams). Higher scores indicate higher consumption of the food item.
National Cancer Institute Dietary Screener Questionnaire Score | Month 12
  27-item self-assessment of frequency of consumption of selected foods and drinks over the past month.
  The scoring procedure converts responses to estimates of individual dietary intake for: Fruits and Vegetables (cup equivalents); Dairy (cup equivalents); Added Sugars (teaspoon equivalents); Whole Grains (ounce equivalents); Fiber (grams); and Calcium (milligrams). Higher scores indicate higher consumption of the food item.
International Physical Activity Questionnaire (IPAQ) Short-Version Score | Baseline
  Self-assessment providing an estimate of the number of minutes per week participants engage in three categories of physical activity: vigorous activity, moderate activity, and walking activity.
  Results are expressed in metabolic equivalent (MET) minutes per week. MET minutes represent the amount of energy expended carrying out physical activity.
  The formula for calculating MET is as follows: 8(vigorous activity)(minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes) = MET.
  Higher scores indicate higher weekly levels of physical activity.
International Physical Activity Questionnaire (IPAQ) Short-Version Score | Month 6
  Self-assessment providing an estimate of the number of minutes per week participants engage in three categories of physical activity: vigorous activity, moderate activity, and walking activity.
  Results are expressed in metabolic equivalent (MET) minutes per week. MET minutes represent the amount of energy expended carrying out physical activity.
  The formula for calculating MET is as follows: 8(vigorous activity)(minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes) = MET.
  Higher scores indicate higher weekly levels of physical activity.
International Physical Activity Questionnaire (IPAQ) Short-Version Score | Month 12
  Self-assessment providing an estimate of the number of minutes per week participants engage in three categories of physical activity: vigorous activity, moderate activity, and walking activity.
  Results are expressed in metabolic equivalent (MET) minutes per week. MET minutes represent the amount of energy expended carrying out physical activity.
  The formula for calculating MET is as follows: 8(vigorous activity)(minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes) = MET.
  Higher scores indicate higher weekly levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hu, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Lu.hu@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Lu.hu@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.